CLINICAL TRIAL: NCT01596062
Title: Prospective, Multicenter, Randomized, Open-label, Phase 2, Lasting 12 Weeks, Evaluating the Pharmacodynamics, Efficacy and Safety of Basiliximab in de Novo Adult Renal Transplant Patients at Low Risk Receiving Either a Cumulative Dose of Basiliximab of 40 or 80 mg in Combination With Cyclosporine Microemulsion, or a Cumulative Dose of 80 mg of Basiliximab Without Calcineurin Inhibitor, With Additional Follow-up of 12 Weeks
Brief Title: Pharmacodynamics, Efficacy and Safety of Basiliximab 40 or 80 mg in Combination With Ciclosporine Microemulsion or Everolimus, in Adult Low Risk de Novo Renal Transplant Recipients (IDEALE Study)
Acronym: IDEALE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCHI621AFR05; 2010-024231-16 (EudraCT Number); NCT01469390 (obsolete NCT alias)
Record Dates: First submitted 2011-09-29; First posted 2012-05-10 (Estimated); Results first posted 2014-07-25 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-06

CONDITIONS: Renal Transplantation
Keywords: Basiliximab; renal transplantation; CNI-free; everolimus
MeSH Terms: interventions — Basiliximab; Cyclosporine; Everolimus; Mycophenolic Acid; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Simulect 40mg + Neoral + Myfortic + steroids (Active Comparator): A cumulative dose of 40 mg of Simulect® (20mg at Day 0 (D0) and 20mg at Day 4 (D4)+ Neoral® + Myfortic® + corticosteroids
  Interventions: Drug: Simulect®; Drug: Neoral®; Drug: Myfortic®; Drug: Corticosteroids
- Simulect 80mg + Neoral + Myfortic + steroids (Experimental): A cumulative dose of 80 mg of Simulect® (40mg at D0 and 40mg at D4) + Neoral® + Myfortic® + corticosteroids
  Interventions: Drug: Simulect®; Drug: Neoral®; Drug: Myfortic®; Drug: Corticosteroids
- Simulect 80mg + Certican + Myfortic + steroids (Experimental): A cumulative dose of 80 mg of Simulect® (40mg at D0 and 40mg at D4) + Certican® + Myfortic® + corticosteroids
  Interventions: Drug: Simulect®; Drug: Certican®; Drug: Myfortic®; Drug: Corticosteroids

INTERVENTIONS:
Drug: Simulect® — Simulect® was provided to the study center in its commercial package containing a powder vial with 20 mg of active product and sterile water for injection. The solution should be used immediately after reconstitution. The infusion was prepared by adding at least 50 mL of physiologic or 5% glucose solution to the reconstituted solution (at least 100 mL for 40 mg of Simulect®). Simulect® was transported and kept in a cold environment (2-8°C) as recommended in the summary of product characteristics (SPC).
  Other Names: Basiliximab
Drug: Neoral® — Neoral® was provided to the study center in its commercial package as 10, 25, 50 or 100 mg soft capsules in thermoformed blister packs.
  Other Names: Cyclosporine microemulsion
  Arms: Simulect 40mg + Neoral + Myfortic + steroids; Simulect 80mg + Neoral + Myfortic + steroids
Drug: Certican® — Certican® was provided to the study center in its commercial package as 0.75, 0.5 and 0.25 mg tablets in thermoformed blister packs.
  Other Names: Everolimus
  Arms: Simulect 80mg + Certican + Myfortic + steroids
Drug: Myfortic® — Myfortic® was administered orally b.i.d. with a 12-hour interval. Tablets could be taken either with or outside meals but consistently throughout the study. To maintain the integrity of the enteric coating, tablets were not to be crushed. Myfortic® treatment was initiated either preoperatively or within 24 hours post transplantation according to local practice in each center. Starting dose was to be 2160 mg/day (1080 mg b.i.d.) for at least 2 weeks and for at most 4 weeks. Patients were then to receive 1440 mg/day (720 mg b.i.d.) until the end of the study. Myfortic® was administered as concomitant treatment to all patients, using the same regimen for all 3 study groups. It was provided to the study center in its commercial package as 180 and 360 mg gastro-resistant tablets.
  Other Names: mycophenolate sodium
Drug: Corticosteroids — Corticosteroid i.v. therapy could be administered peri or per operatively according to local practice in each center with the same scheme for each patient in the center. Oral corticotherapy was to be initiated rapidly, within one week following transplantation, with a minimal dose of 20 mg/day. Thereafter, the dose was to be decreased according to local practice but oral corticosteroids were to be continued throughout the study with a minimal dose of 5 mg/day.

SUMMARY:
The aims of this study are to extensively study the levels of CD25-Receptors saturation and expression obtained with 2 different doses of Simulect® in combination with Neoral® (i.e to demonstrate that saturation and expression vary according to the dose of Simulect® given), and to study the levels of CD25-Receptors saturation without Neoral® and compare them to the data with Neoral®.

It will be conducted in low risk de novo adult renal transplant recipients until 12 weeks post-transplant, receiving either a cumulative dose of 40 or 80 mg of Simulect® in combination with Neoral®, or a cumulative dose of 80 mg of Simulect® in a calcineurin inhibitor free immunosuppressant therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving a primary renal graft from a deceased or living, related or unrelated donor and who require basiliximab induction therapy
* Cold ischemia time < 30 hours

Exclusion (Non inclusion) criteria:

* Patients undergoing multi-organ transplantation, including both kidneys, or who have previously undergone organ transplantation, including renal transplantation
* Patients receiving a graft from a non-heart-beating donor
* A-B-O incompatible graft or positive T cell crossmatch
* Patients receiving a graft from an expanded criteria donor according to the UNOS definition (donor older than 60 years or donor aged between 50 and 60 years and presence of at least 2 of the following factors: hypertension, serum creatinine concentration ≥ 132 µmol/mL, cardiovascular cause of death)
* Positive anti-HLA antibodies (Luminex) prior to transplantation
* Patients whose original renal disease was primary focal and segmental hyalinosis or was related to atypical hemolytic uremic syndrome
* EBV-negative patients receiving a graft from an EBV-positive donor (EBV D+R-)

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- France (3):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Tours

REFERENCES:
- [Derived] Thibault G, Paintaud G, Legendre C, Merville P, Coulon M, Chasseuil E, Ternant D, Rostaing L, Durrbach A, Di Giambattista F, Buchler M, Lebranchu Y. CD25 blockade in kidney transplant patients randomized to standard-dose or high-dose basiliximab with cyclosporine, or high-dose basiliximab in a calcineurin inhibitor-free regimen. Transpl Int. 2016 Feb;29(2):184-95. doi: 10.1111/tri.12688. Epub 2015 Oct 8. PMID 26369526

RESULTS

PARTICIPANT FLOW:
Recruitment Details: With premature end of recruitment only 16 patients were included. Descriptive analysis was done & statistical method fitted the small number of patients. One final analysis was performed at M6 post-transplantation & comprised assessment of criteria planned at M3 and M6. Some analysis pertaining to the secondary objectives were not performed.
Period: Overall Study
Arm/Group | Simulect 40mg + Neoral + Myfortic + Steroids | Simulect 80mg + Neoral + Myfortic + Steroids | Simulect 80mg + Certican + Myfortic + Steroids
Started | 3 | 6 | 7
Completed | 2 | 6 | 4
Not Completed | 1 | 0 | 3
Not completed — Adverse Event | 1 | 0 | 2
Not completed — Lack of Efficacy | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Simulect 40mg + Neoral + Myfortic + Steroids | Simulect 80mg + Neoral + Myfortic + Steroids | Simulect 80mg + Certican + Myfortic + Steroids | Total
Number analyzed (Participants) | 3 | 6 | 7 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (8.7) | 45.0 (11.4) | 39.7 (12.2) | 44.3 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2 | 4
  Male | 3 | 4 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) of CD25 Saturation by Basiliximab From Day 0 to Day 84
Description: CD25 saturation is the percentage of T cells expressing CD25. Mean AUC of CD25 was calculated only for patients who received two Simulect® injections.
Time Frame: Day 84 (Week 12) after transplantation
Population: PK/PD population: Patients included in the ITT population for whom at least one blood sample for PK/PD analyses was collected. This population is the reference population for the PK and PD analyses.
Measure: Mean (Standard Deviation); unit: Weeks * Percentage of saturated CD25
Arm/Group | Simulect 40mg + Neoral + Myfortic + Steroids | Simulect 80mg + Neoral + Myfortic + Steroids | Simulect 80mg + Certican + Myfortic + Steroids
Number analyzed (Participants) | 3 | 6 | 6
Weeks * Percentage of saturated CD25 | 8.4 (1.61) | 11.1 (1.12) | 9.7 (0.70)

2. Primary Outcome: Saturation Rate of CD25 Antigen Saturation by Basiliximab
Description: CD25 saturation is the percentage of T cells expressing CD25
Time Frame: Day 0, Day 1, Day 4, Day 6, Day 14, Day 21, Day 28, Day 42, Day 56 and Day 84 (Week 12) post-transplantation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of T cells
Arm/Group | Simulect 40mg + Neoral + Myfortic + Steroids | Simulect 80mg + Neoral + Myfortic + Steroids | Simulect 80mg + Certican + Myfortic + Steroids
Number analyzed (Participants) | 3 | 6 | 7
percentage of T cells
  Day 0 (before injection) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Day 0 (2 hours after injection) | 93.7 (10.97) | 96.7 (8.16) | 94.7 (5.19)
  Day 1 | 95.7 (7.51) | 97.7 (5.24) | 99.0 (2.65)
  Day 4 (before injection); (n= 3, 6, 6) | 100.0 (0.00) | 96.2 (6.88) | 93.7 (9.89)
  Day 4 (2 hours after injection): (n= 3, 6, 5) | 96.7 (5.77) | 96.3 (6.83) | 84.8 (19.25)
  Day 6: (n= 3, 6, 6) | 98.7 (2.31) | 100.0 (0.00) | 94.0 (14.70)
  Day 14: (n= 3, 6, 6) | 98.3 (2.89) | 96.7 (7.23) | 97.3 (6.53)
  Day 21: (n= 3, 6, 6) | 100.0 (0.00) | 94.5 (10.80) | 92.5 (11.83)
  Day 28: (n= 3, 6, 6) | 95.3 (4.16) | 100.0 (0.00) | 92.7 (9.33)
  Day 42: (n= 3, 6, 5) | 78.3 (9.07) | 100.0 (0.00) | 99.2 (1.79)
  Day 56: (n= 3, 6, 5) | 65.0 (56.35) | 93.3 (13.20) | 94.2 (12.97)
  Day 84 (Week 12): (n= 3, 6, 5) | 0.0 (0.00) | 67.5 (48.55) | 14.2 (20.86)

3. Secondary Outcome: AUC of Basiliximab Binding to CD25 Receptors From Day 0 to Day 84
Description: Mean AUC was calculated only for patients who received two Simulect injections.
Time Frame: Day 84 (Week 12) post-transplantation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Weeks * Percentage of T cells
Arm/Group | Simulect 40mg + Neoral + Myfortic + Steroids | Simulect 80mg + Neoral + Myfortic + Steroids | Simulect 80mg + Certican + Myfortic + Steroids
Number analyzed (Participants) | 3 | 6 | 6
Weeks * Percentage of T cells | 7.0 (1.80) | 9.9 (2.22) | 8.4 (0.75)

4. Secondary Outcome: Percentage of T-cells That Bind Basiliximab to CD25 Receptors
Description: This is the percentage of T cells binding basiliximab at all timepoints.
Time Frame: Day 0, Day 1, Day 4, Day 6, Day 14, Day 21, Day 28, Day 42, Day 56 and Day 84 (Week 12) post-transplantation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of T cells
Arm/Group | Simulect 40mg + Neoral + Myfortic + Steroids | Simulect 80mg + Neoral + Myfortic + Steroids | Simulect 80mg + Certican + Myfortic + Steroids
Number analyzed (Participants) | 3 | 6 | 7
Percentage of T cells
  Day 0 (before injection) | 0.0 (0.00) | 0.0 (0.00) | 4.7 (12.47)
  Day 0 (2 hours after injection) | 95.3 (8.08) | 96.2 (9.39) | 81.6 (28.30)
  Day 1 (n= 3, 5, 7) | 70.0 (28.58) | 64.8 (35.15) | 91.4 (11.65)
  Day 4 (before injection): (n= 3, 6, 6) | 100.0 (0.00) | 59.0 (45.98) | 53.0 (33.33)
  Day 4 (2 hours after injection): (n= 3, 5, 5) | 100.0 (0.00) | 83.4 (20.14) | 81.2 (16.02)
  Day 6: (n= 3, 6, 6) | 91.7 (14.43) | 99.0 (2.45) | 98.3 (4.08)
  Day 14: (n= 3, 6, 6) | 100.0 (0.00) | 89.0 (22.00) | 93.8 (15.11)
  Day 21: (n= 3, 6, 6) | 89.0 (19.05) | 87.7 (26.93) | 85.8 (32.31)
  Day 28: (n= 3, 6, 6) | 76.3 (17.62) | 91.0 (14.00) | 82.7 (26.29)
  Day 42: (n= 3, 6, 5) | 47.3 (28.22) | 84.0 (19.75) | 78.8 (30.11)
  Day 56: (n= 3, 6, 5) | 53.0 (41.80) | 88.8 (27.35) | 75.2 (15.29)
  Day 84 (Week 12): (n= 3, 6, 5) | 6.7 (6.11) | 57.7 (43.83) | 15.8 (9.73)

5. Secondary Outcome: Proportion of CD3+, CD4+, CD8+, CD19+ and CD56+ T Cells
Description: Cell counts of various subpopulations of T, B and NK lymphocytes (CD3, CD4, CD8, CD19 and CD56) (flow cytometry).
Time Frame: Day 0, Day 6, Day 42, Day 84 (Week 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Simulect 40mg + Neoral + Myfortic + Steroids | Simulect 80mg + Neoral + Myfortic + Steroids | Simulect 80mg + Certican + Myfortic + Steroids
Number analyzed (Participants) | 3 | 6 | 7
10^9 cells/L
  CD3 cells count at Day 0 (before injection) | 0.5 (0.25) | 0.9 (0.28) | 0.7 (0.28)
  CD3 cells count at Day 6: (n= 3, 6, 6) | 0.6 (0.39) | 1.1 (0.50) | 0.9 (0.75)
  CD3 cells count at Day 42: (n= 3, 6, 5) | 0.5 (0.09) | 1.2 (0.96) | 1.1 (1.18)
  CD3 cells count at Day 84 (Week 12): (n= 3, 6, 6) | 0.8 (0.58) | 1.2 (0.72) | 1.1 (1.22)
  CD4 cells count at Day 0 (before injection) | 0.4 (0.19) | 0.6 (0.20) | 0.5 (0.22)
  CD4 cells count at Day 6: (n= 3, 6, 6) | 0.5 (0.30) | 0.7 (0.28) | 0.6 (0.59)
  CD4 cells count at Day 42: (n= 3, 6, 5) | 0.3 (0.08) | 0.8 (0.53) | 0.8 (0.82)
  CD4 cells count at Day 84 (Week 12): (n= 3, 6, 6) | 0.6 (0.36) | 0.8 (0.42) | 0.7 (0.86)
  CD8 cells count at Day 0 (before injection) | 0.1 (0.05) | 0.3 (0.13) | 0.2 (0.15)
  CD8 cells count at Day 6: (n= 3, 6, 6) | 0.2 (0.08) | 0.3 (0.25) | 0.2 (0.24)
  CD8 cells count at Day 42: (n= 3, 6, 5) | 0.1 (0.05) | 0.3 (0.44) | 0.4 (0.37)
  CD8 cells count at Day 84 (Week 12): (n= 3, 6, 6) | 0.2 (0.24) | 0.3 (0.32) | 0.3 (0.37)
  CD19 cells count at Day 0 (before injection) | 0.1 (0.08) | 0.1 (0.10) | 0.1 (0.05)
  CD19 cells count at Day 6: (n=3, 6, 6) | 0.1 (0.07) | 0.2 (0.27) | 0.2 (0.17)
  CD19 cells count at Day 42: (n= 3, 6, 5) | 0.1 (0.09) | 0.2 (0.21) | 0.2 (0.18)
  CD19 cells count at Day 84 (Week 12): (n= 3, 6, 6) | 0.2 (0.20) | 0.1 (0.11) | 0.1 (0.15)
  CD56 cells count at Day 0 (before injection) | 0.1 (0.20) | 0.2 (0.14) | 0.2 (0.31)
  CD56 cells count at Day 6: (n= 3, 6, 6) | 0.1 (0.00) | 0.1 (0.06) | 0.2 (0.25)
  CD56 cells count at Day 42: (n= 3, 6, 5) | 0.1 (0.05) | 0.2 (0.10) | 0.2 (0.13)
  CD56 cells count at Day 84 (Week 12): (n= 3, 6, 6) | 0.1 (0.05) | 0.1 (0.03) | 0.1 (0.15)

6. Secondary Outcome: Percentage of Participants With of Biopsy Proven Acute Rejection (BPAR)
Description: BPAR is one of the components of treatment failure. One assessment of efficacy was BPAR. Renal graft biopsies were performed and the renal tissue was examined to determine if there was acute rejection of the renal transplant.
Time Frame: Day 84 (Week 12), Week 24 post-transplantation
Population: Intent to treat (ITT) population: All randomized patients having received at least one Simulect® injection and who had been transplanted. This population is the reference population for the efficacy analyses.
Measure: Number; unit: Percentage of participants
Arm/Group | Simulect 40mg + Neoral + Myfortic + Steroids | Simulect 80mg + Neoral + Myfortic + Steroids | Simulect 80mg + Certican + Myfortic + Steroids
Number analyzed (Participants) | 3 | 6 | 7
Percentage of participants
  Day 84 (Week 12): No | 66.7 | 83.3 | 42.9
  Day 84 (Week 12):Yes | 33.3 | 16.7 | 57.1
  Week 24: No | 66.7 | 83.3 | 42.9
  Week 24:Yes | 33.3 | 16.7 | 57.1

7. Secondary Outcome: Percentage of Participants With Biopsy Proven Acute Rejection (BPAR) According to Type and Severity
Description: Antibody mediated acute rejection: C4d deposition, presence of circulating antidonor antibody, morphologic evidence of acute tissue injury such as acute tubular necrosis-like minimal inflammation or capillary and/or glomerular inflammation and/or thromboses or arterial inflammation. Cellular acute rejection: acute T-cell mediated rejection Type IA: Significant interstitial infiltration (> 25% of parenchyma) and foci of moderate tubulitis (> 4 mononuclear cells/tubular cross section or group of 10 tubular cells) Type IB: Significant interstitial infiltration (> 25% of parenchyma) and foci of severe tubulitis (> 10 mononuclear cells/tubular cross section or group of 10 tubular cells) Type IIA: Mild to moderate intimal arteritis. Type IIB: Severe intimal arteritis comprising > 25% of the lumenal area. Type III: Transmural (full vessel wall thickness) arteritis and/or arterial fibrinoid change and necrosis of medial smooth muscle cells (with accompanying lymphocytic inflammation).
Time Frame: Day 84 (Week 12), Week 24 post-transplantation
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Simulect 40mg + Neoral + Myfortic + Steroids | Simulect 80mg + Neoral + Myfortic + Steroids | Simulect 80mg + Certican + Myfortic + Steroids
Number analyzed (Participants) | 3 | 6 | 7
Percentage of participants
  Day 84 (Week 12): Antibody mediated AR - No | 66.7 | 100.0 | 85.7
  Day 84 (Week 12): Antibody mediated AR - Yes | 33.3 | 0.0 | 14.3
  Day 84 (Week 12): Cellular AR - No | 100.0 | 83.3 | 57.1
  Day 84 (Week 12): Cellular AR - Yes | 0.0 | 16.7 | 42.9
  Day 84 (Week 12): Banff type lA | 0.0 | 0.0 | 14.3
  Day 84 (Week 12): Banff type lB | 0.0 | 16.7 | 14.3
  Day 84 (Week 12): Banff type llA | 0.0 | 0.0 | 0.0
  Day 84 (Week 12): Banff type llB | 0.0 | 0.0 | 14.3
  Day 84 (Week 12): Banff type lll (C AR) | 0.0 | 0.0 | 0.0
  Week 24: Antibody mediated AR - No | 66.7 | 100.0 | 85.7
  Week 24: Antibody mediated AR - Yes | 33.3 | 0.0 | 14.3
  Week 24: Cellular AR - No | 100.0 | 83.3 | 57.1
  Week 24: Cellular AR - Yes | 0.0 | 16.7 | 42.9
  Week 24: Banff type lA | 0.0 | 0.0 | 0.0
  Week 24: Banff type lB | 0.0 | 16.7 | 28.6
  Week 24: Banff type llA | 0.0 | 0.0 | 0.0
  Week 24: Banff type llB | 0.0 | 0.0 | 14.3
  Week 24: Banff type lll | 0.0 | 0.0 | 0.0

8. Secondary Outcome: Percentage of Participants With of Treatment Failures
Description: Treatment failure was defined either as a BPAR, a graft loss, a death or a loss to follow-up. An extended treatment failure was also defined including treated borderline lesions, BPAR, graft loss, death or loss to follow-up. Treated borderline lesions were considered as acute rejection by investigators and DMC experts.
Time Frame: Day 84 (Week 12), Week 24
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Simulect 40mg + Neoral + Myfortic + Steroids | Simulect 80mg + Neoral + Myfortic + Steroids | Simulect 80mg + Certican + Myfortic + Steroids
Number analyzed (Participants) | 3 | 6 | 7
Percentage of participants
  Day84 (Week 12): BPAR and/or borderline lesions-No | 66.7 | 66.7 | 14.3
  Day84 (Week 12):BPAR and/or borderline lesions-Yes | 33.3 | 33.3 | 85.7
  Day 84 (Week 12): Graft loss - No | 66.7 | 100.0 | 100.0
  Day 84 (Week 12): Graft loss - Yes | 33.3 | 0.0 | 0.0
  Day 84 (Week 12): Death - No | 100.0 | 100.0 | 100.0
  Day 84 (Week 12): Death - Yes | 0.0 | 0.0 | 0.0
  Day 84 (Week 12): Loss to follow-up - No | 100.0 | 100.0 | 100.0
  Day 84 (Week 12): Loss to follow-up - Yes | 0.0 | 0.0 | 0.0
  Week 24: BPAR or borderline lesions - No | 66.7 | 66.7 | 14.3
  Week 24: Graft loss - No | 66.7 | 100.0 | 100.0
  Week 24: Death - No | 100.0 | 100.0 | 100.0
  Week 24: Loss to follow-up - No | 100.0 | 100.0 | 100.0
  Week 24: Loss to follow-up - Yes | 0.0 | 0.0 | 0.0
  Week 24: BPAR or borderline lesions - Yes | 33.3 | 33.3 | 85.7
  Week 24: Graft loss - Yes | 33.3 | 0.0 | 0.0
  Week 24: Death - Yes | 0.0 | 0.0 | 0.0

9. Secondary Outcome: Estimated Glomerular Filtration Rate (eGFR) at Day 8 and Week 24
Description: (MDRDa formula) with imputation by last observation carried forward (LOCF)
Time Frame: Day 8, Week 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Simulect 40mg + Neoral + Myfortic + Steroids | Simulect 80mg + Neoral + Myfortic + Steroids | Simulect 80mg + Certican + Myfortic + Steroids
Number analyzed (Participants) | 3 | 6 | 7
mL/min/1.73m^2
  Day 8 | 35.0 (13.20) | 53.8 (23.79) | 49.9 (18.45)
  Week 24 (n= 3, 6, 6) | 31.9 (27.93) | 55.7 (15.68) | 54.4 (10.48)

ADVERSE EVENTS:
Arm/Group | Simulect 40mg + Neoral + Myfortic + Steroids | Simulect 80mg + Neoral + Myfortic + Steroids | Simulect 80mg + Certican + Myfortic + Steroids
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/6 | 5/7
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Simulect 40mg + Neoral + Myfortic + Steroids (N=3) | Simulect 80mg + Neoral + Myfortic + Steroids (N=6) | Simulect 80mg + Certican + Myfortic + Steroids (N=7)
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Kidney transplant rejection (Immune system disorders) | 0 | 0 | 1
Transplant rejection (Immune system disorders) | 1 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Graft loss (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 2
Epididymitis (Reproductive system and breast disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Lymphocele (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Simulect 40mg + Neoral + Myfortic + Steroids (N=3) | Simulect 80mg + Neoral + Myfortic + Steroids (N=6) | Simulect 80mg + Certican + Myfortic + Steroids (N=7)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 2
Ascites (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Gingival hypertrophy (Gastrointestinal disorders) | 1 | 1 | 0
Lip pruritus (Gastrointestinal disorders) | 0 | 1 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 1
Oedema (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 3 | 1 | 1
Cholestasis (Hepatobiliary disorders) | 1 | 0 | 0
Cytolytic hepatitis (Hepatobiliary disorders) | 1 | 3 | 0
BK virus infection (Infections and infestations) | 0 | 0 | 1
Gingival infection (Infections and infestations) | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 1 | 0
Otitis media (Infections and infestations) | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 | 0 | 1
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 1 | 0 | 1
Incision site pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 1
Weight increased (Investigations) | 1 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 0 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Hirsutism (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 2 | 1 | 4
Intra-abdominal haematoma (Vascular disorders) | 0 | 0 | 2
Phlebitis superficial (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.